CLINICAL TRIAL: NCT02320058
Title: A Multi-Center Phase 2 Open-Label Study to Evaluate Safety and Efficacy in Subjects With Melanoma Metastatic to the Brain Treated With Nivolumab in Combination With Ipilimumab Followed by Nivolumab Monotherapy
Brief Title: An Investigational Immuno-therapy Study to Evaluate Safety and Effectiveness in Patients With Melanoma That Has Spread to the Brain, Treated With Nivolumab in Combination With Ipilimumab, Followed by Nivolumab by Itself
Acronym: CheckMate204
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-204
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and Ipilimumab (Experimental): Induction Phase: Nivolumab + Ipilimumab infusion intravenously
  Maintenance Phase: Nivolumab infusion intravenously
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: Yervoy
Drug: Nivolumab
  Other Names: Opdivo; BMS-936558

SUMMARY:
This is a study of Nivolumab combined with Ipilimumab followed by Nivolumab by itself for the treatment of patients with Melanoma that has spread to the brain. Patients with histologically confirmed Malignant Melanoma and asymptomatic brain metastases are eligible for the study.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

1. Target Population

1. Histologically confirmed malignant melanoma with measurable metastases in the brain. Both asymptomatic and symptomatic patients.
2. Cohort A (asymptomatic patients): At least 1 measurable brain metastasis ≥ 0.5 cm in and ≤ 3 cm in longest diameter that has not been previously irradiated. No clinical requirement for local intervention (surgery, radiosurgery, corticosteroid therapy) or other systemic therapy

   Cohort B (symptomatic patients): Subjects with neurologic signs and symptoms related to metastatic brain lesions are eligibile. Subjects must have at least 1 measurable brain metastasis ≥ 0.5 cm in and ≤ 3 cm in longest diameter that has not been previously irradiated. No immediate requirement (within 3 weeks prior to first treatment) for local intervention (surgery, radiosurgery, corticosteroid therapy). Steroid use is permitted as defined in the protocol.
3. Prior stereotactic radiotherapy (SRT) and prior excision of up to 3 melanoma brain metastases is permitted if there has been complete recovery, with no neurologic sequelae, and measurable lesions remain. Growth or change in a lesion previously irradiated will not be considered measurable. Regrowth in cavity of previously excised lesion will not be considered measurable. lesions or prior excision must have occurred ≥ 3 weeks before the start of dosing for this study
4. Must have tumor tissue available for biomarker analysis. Biopsy should be excisional, incisional, punch, or core needle
5. Cohort A (asymptomatic): Subjects must be free of neurologic signs and symptoms related to metastatic brain lesions and must not have required or received systemic corticosteroid therapy within 10 days prior to first treatment.

   Cohort B (symptomatic): Subjects with neurologic signs and symptoms related to metastatic brain lesions are eligible per Amendment 02. Subjects with neurologic signs and symptoms may be treated with a total daily dose of no more than 4 mg of dexamethasone that is stable or tapering for 10 days prior to first treatment. Subjects with neurologic signs and symptoms who are not being treated with steroids are eligible for Cohort B and should have no experience of seizure within 10 days prior to first treatment.
6. Allowable prior therapy:

   1. Approved adjuvant therapies, which may include molecularly-targeted agents, IFN α, and ipilimumab. Patients who received ipilimumab as adjuvant therapy must have a 6 month washout before receiving any dosing on this study
   2. For advanced disease, interleukin-2 at any dose and/or IFN-α (any formulation, no washout required); MEK and BRAF inhibitors: washout for at least 4 weeks prior to the start of dosing in this study
   3. Steroids for physiological replacement are allowed.
7. Cohort A (asymptomatic): ECOG performance status ≤1 Cohort B (symptomatic): ECOG performance status ≤2

Exclusion Criteria:

2. Target Disease Exceptions

1. History of known leptomeningeal involvement (lumbar puncture not required)
2. Previous stereotactic or highly conformal radiotherapy within 3 weeks before the start of dosing for this study. Note the stereotactic radiotherapy field must not have included the brain index lesion(s)
3. Brain lesions >3 lesions which were previously treated with SRT
4. Brain lesion size > 3cm 3. Medical History and Concurrent Diseases

a) History of whole brain irradiation b) Subjects with an active, known or suspected autoimmune disease c) Subjects with major medical, neurologic or psychiatric condition who are judged as unable to fully comply with study therapy or assessments should not be enrolled d) Any concurrent malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix. For any prior invasive malignancy, at least 5 years must have elapsed since curative therapy and patients must have no residual sequelae of prior therapy e) Cohort A (asymptomatic): The use of corticosteroids is not allowed within 10 days prior to first treatment (based upon 5 times the expected half life of dexamethasone) except patients who are taking steroids for physiological replacement. If alternative corticosteroid therapy has been used, consultation with the sponsor Medical Monitor is required to determine the washout period prior to initiating study treatment Cohort B (symptomatic): Subjects with neurologic sign and symptoms related to brain metastases who are being treated with a total daily dose of higher than 4 mg dexamethasone or equivalent within 10 prior to the start of treatment with study drug are excluded.

4. Physical and Laboratory Test Findings

1. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
2. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) even if fully immunocompetent on ART-due to the unknown effects of HIV on the immune response to combined nivolumab plus ipilimumab or the unique toxicity spectrum of these drugs in patients with HIV

   5. Allergies and Adverse Drug Reaction

a) History of allergy to study drug components b) History of severe hypersensitivity reaction to any monoclonal antibody

6. Other Exclusion Criteria

1. Prisoners or subjects who are involuntarily incarcerated
2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness Eligibility criteria for this study have been carefully considered to ensure the safety of the study subjects and that the results of the study can be used. It is imperative that subjects fully meet all eligibility criteria

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (36):
- United States (36):
  - City of Hope, Duarte, California
  - Angeles Clinic and Research Institute, Los Angeles, California
  - UCLA Medical Hematology and Oncology, Los Angeles, California
  - Stanford University, Palo Alto, California
  - The California Pacific Medical Research Institute, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado - Cancer Center - PPDS, Aurora, Colorado
  - Washington Cancer Inst at MedStar Washington Hospital Ctr, Washington D.C., District of Columbia
  - Weinberg Cancer Institute At Franklin Square, Washington D.C., District of Columbia
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Medical Center, Miami Beach, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - The Cleveland Clinic Foundation, Weston, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case School of Medicine University Hospitals of Cleveland, Cleveland, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - St Luke's Health Network, Easton, Pennsylvania
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute - PPDS, Salt Lake City, Utah
  - Inova Melanoma and Skin Cancer Center, Fairfax, Virginia

REFERENCES:
- [Derived] Huang RY, Youssef G, Nelson T, Wen PY, Forsyth P, Hodi FS, Margolin K, Algazi AP, Hamid O, Lao CD, Ernstoff MS, Moschos SJ, Atkins MB, Postow MA, Reardon DA, Grootendorst DJ, Leung D, Askelson M, Ritchings C, Tawbi HA. Comparative Analysis of Intracranial Response Assessment Criteria in Patients With Melanoma Brain Metastases Treated With Combination Nivolumab + Ipilimumab in CheckMate 204. J Clin Oncol. 2025 Apr;43(10):1210-1218. doi: 10.1200/JCO.24.00953. Epub 2025 Jan 3. PMID 39752606
- [Derived] Johannet P, Simons M, Qian Y, Azmy N, Mehnert JM, Weber JS, Zhong J, Osman I. Risk and tropism of central nervous system (CNS) metastases in patients with stage II and III cutaneous melanoma. Cancer. 2022 Oct;128(20):3620-3629. doi: 10.1002/cncr.34435. Epub 2022 Aug 25. PMID 36006879
- [Derived] Tawbi HA, Forsyth PA, Hodi FS, Algazi AP, Hamid O, Lao CD, Moschos SJ, Atkins MB, Lewis K, Postow MA, Thomas RP, Glaspy J, Jang S, Khushalani NI, Pavlick AC, Ernstoff MS, Reardon DA, Kudchadkar R, Tarhini A, Chung C, Ritchings C, Durani P, Askelson M, Puzanov I, Margolin KA. Long-term outcomes of patients with active melanoma brain metastases treated with combination nivolumab plus ipilimumab (CheckMate 204): final results of an open-label, multicentre, phase 2 study. Lancet Oncol. 2021 Dec;22(12):1692-1704. doi: 10.1016/S1470-2045(21)00545-3. Epub 2021 Nov 10. PMID 34774225
- [Derived] Tawbi HA, Forsyth PA, Hodi FS, Lao CD, Moschos SJ, Hamid O, Atkins MB, Lewis K, Thomas RP, Glaspy JA, Jang S, Algazi AP, Khushalani NI, Postow MA, Pavlick AC, Ernstoff MS, Reardon DA, Puzanov I, Kudchadkar RR, Tarhini AA, Sumbul A, Rizzo JI, Margolin KA. Safety and efficacy of the combination of nivolumab plus ipilimumab in patients with melanoma and asymptomatic or symptomatic brain metastases (CheckMate 204). Neuro Oncol. 2021 Nov 2;23(11):1961-1973. doi: 10.1093/neuonc/noab094. PMID 33880555
- [Derived] Tawbi HA, Forsyth PA, Algazi A, Hamid O, Hodi FS, Moschos SJ, Khushalani NI, Lewis K, Lao CD, Postow MA, Atkins MB, Ernstoff MS, Reardon DA, Puzanov I, Kudchadkar RR, Thomas RP, Tarhini A, Pavlick AC, Jiang J, Avila A, Demelo S, Margolin K. Combined Nivolumab and Ipilimumab in Melanoma Metastatic to the Brain. N Engl J Med. 2018 Aug 23;379(8):722-730. doi: 10.1056/NEJMoa1805453. PMID 30134131
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 119 participants treated
Groups:
- Cohort A: Asymptomatic patients treated with Nivolumab IV 1 mg/kg Q3W + Ipilimumab IV 3 mg/kg Q3W for a total of 4 doses of the combination therapy followed by Nivolumab IV 3 mg/kg BID for a maximum of 24 months or until progression or until unacceptable toxicity.
- Cohort B: Symptomatic patients treated with Nivolumab IV 1 mg/kg Q3W + Ipilimumab IV 3 mg/kg Q3W for a total of 4 doses of the combination therapy followed by Nivolumab IV 3 mg/kg BID for a maximum of 24 months or until progression or until unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 101 | 18
Completed | 59 | 5
Not Completed | 42 | 13
Not completed — Death | 25 | 10
Not completed — Lost to Follow-up | 4 | 0
Not completed — Other reasons | 4 | 1
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Not reported | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 101 | 18 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (12.29) | 58.2 (13.24) | 58.0 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 5 | 38
  Male | 68 | 13 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 99 | 15 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 99 | 17 | 116
  Black or African American | 0 | 0 | 0
  Asian | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Clinical Benefit Rate (CBR)
Description: Intracranial Clinical Benefit Rate (CBR) is defined as the percentage of all treated participants whose best overall response is either a complete response (CR) or partial response (PR) or whose best overall response was Stable Disease (SD) with duration of >6 months, as determined by modified RECIST 1.1 criteria for index intracranial lesions based on investigator review.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Percentage of Participants | 57.4 [47.2 to 67.2] | 16.7 [3.6 to 41.4]

2. Secondary Outcome: Intracranial Objective Response Rate (ORR)
Description: Investigator-Assessed Intracranial Objective Response Rate (ORR) per modified RECIST 1.1 criteria is defined as the number of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of treated participants.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Percentage of Participants | 53.5 [43.3 to 63.5] | 16.7 [3.6 to 41.4]

3. Secondary Outcome: Intracranial Progression Free Survival (PFS)
Description: Intracranial progression-free survival (PFS) per modified RECIST 1.1 criteria is defined as the time between the date of first dose of study drug and the first date of documented progression, as determined by the investigator, or death due to any cause, whichever occurs first. Participant who die without a reported progression will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die will be censored on the date of first dose of study drug. Participants who started anti-cancer therapy without a prior reported progression will be censored on the date of their last evaluable tumor assessment prior to the initiation of subsequent anti-cancer therapy.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Months | NA [6.87 to NA] — Median and Upper Limit not reached per the Kaplan-Meier method, as the probability of survival was still above 50% | 1.18 [0.72 to 1.25]

4. Secondary Outcome: Extracranial Clinical Benefit Rate (CBR)
Description: Extracranial Clinical Benefit Rate (CBR) is defined as the percentage of all treated participants whose best overall response is either a complete response (CR) or partial response (PR) or whose best overall response was Stable Disease (SD) with duration of >6 months, as determined by RECIST 1.1 criteria for index extracranial lesions based on investigator review.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Percentage of Participants | 53.5 [43.3 to 63.5] | 22.2 [6.4 to 47.6]

5. Secondary Outcome: Extracranial Objective Response Rate (ORR)
Description: Extracranial Objective Response Rate (ORR) per RECIST 1.1 criteria is defined as the number of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of treated participants.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Percentage of Participants | 48.5 [38.4 to 58.7] | 22.2 [6.4 to 47.6]

6. Secondary Outcome: Extracranial Progression Free Survival (PFS)
Description: Extracranial progression-free survival (PFS) per RECIST 1.1 criteria is defined as the time between the date of first dose of study drug and the first date of documented progression, as determined by the investigator, or death due to any cause, whichever occurs first. Participant who die without a reported progression will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die will be censored on the date of first dose of study drug. Participants who started anti-cancer therapy without a prior reported progression will be censored on the date of their last evaluable tumor assessment prior to the initiation of subsequent anti-cancer therapy.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Months | 39.29 [16.13 to 45.80] | 1.77 [0.79 to NA] — upper limit of the confidence interval is not yet reached

7. Secondary Outcome: Global Clinical Benefit Rate (CBR)
Description: Investigator-assessed global (intracranial + extracranial) clinical benefit rate (CBR) per a combination of modified RECIST 1.1 criteria for intracranial lesions and RECIST 1.1 for extracranial disease is defined as the percentage of all treated participants whose best overall response is either a complete response (CR) or partial response (PR) or whose best overall response was Stable Disease (SD) with duration of >6 months
Time Frame: Up to 66 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Percentage of participants | 55.4 [45.2 to 65.3] | 22.2 [6.4 to 47.6]

8. Secondary Outcome: Global Objective Response Rate (ORR)
Description: Investigator-assessed global objective response rate (ORR) per a combination of modified RECIST 1.1 criteria for intracranial lesions and RECIST 1.1 for extracranial disease is defined as the number of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of treated participants.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Percentage of participants | 51.5 [41.3 to 61.6] | 22.2 [6.4 to 47.6]

9. Secondary Outcome: Global Progression Free Survival (PFS)
Description: Investigator-assessed global progression free survival (PFS) per a combination of modified RECIST 1.1 criteria for intracranial lesions and RECIST 1.1 for extracranial disease is defined as the time between the date of first dose of study drug and the first date of documented progression, as determined by the investigator, or death due to any cause, whichever occurs first. Participant who die without a reported progression will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die will be censored on the date of first dose of study drug. Participants who started anti-cancer therapy without a prior reported progression will be censored on the date of their last evaluable tumor assessment prior to the initiation of subsequent anti-cancer therapy.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Months | 29.54 [6.87 to NA] — upper limit of the confidence interval is not yet reached | 1.18 [0.79 to 4.14]

10. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from the date of the start of treatment until the date of death. For participants who have not died, OS will be censored at the recorded last date of participant contact, and participants with a missing recorded last date of contact will be censored at the last date the participant was known to be alive.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Months | 45.80 [45.80 to NA] — upper limit of the confidence interval is not yet reached | 8.77 [1.77 to NA] — upper limit of the confidence interval is not yet reached

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with any grade of adverse events (AEs) and any grade of serious adverse events (SAEs) graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Time Frame: From first dose to 30 days post last dose (Up to 66 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Participants
  Adverse Events (AEs) | 98 | 18
  Serious Adverse Events (SAEs) | 44 | 11

12. Secondary Outcome: Number of Participants Deaths
Description: Number of participants who died due to any cause.
Time Frame: Up to 66 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Participants | 29 | 10

13. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: Number of participants with laboratory abnormalities in specific liver tests based on US conventional units to determine the safety and tolerability of Nivolumab and Daratumumab. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * ALT or AST > 3 x ULN, > 5 x ULN, > 10 x ULN and > 20 x ULN
  * Total bilirubin > 2 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
Time Frame: From first dose to 30 days post last dose (Up to 66 months)
Population: All treated participants with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 96 | 15
Participants
  ALT OR AST > 3XULN | 25 | 1
  ALT OR AST > 5XULN | 16 | 0
  ALT OR AST > 10XULN | 7 | 0
  ALT OR AST > 20XULN | 2 | 0
  TOTAL BILIRUBIN > 2XULN | 3 | 0
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN ONE DAY | 1 | 0
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN 30 DAYS | 1 | 0

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: Number of participants with laboratory abnormalities in specific thyroid tests based on US conventional units to determine the safety and tolerability of Nivolumab and Daratumumab. The number of subjects with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * TSH value > ULN and
  * with baseline TSH value <= ULN
  * with at least one FT3/FT4 test value < LLN within 2-week window after the abnormal TSH test
  * with all FT3/FT4 test values >= LLN within 2-week window after the abnormal TSH test
  * with FT3/FT4 missing within 2-week window after the abnormal TSH test.
  * TSH < LLN and
  * with baseline TSH value >= LLN
  * with at least one FT3/FT4 test value > ULN within 2-week window after the abnormal TSH test
  * with all FT3/FT4 test values <= ULN within 2-week window after the abnormal TSH test
  * with FT3/FT4 missing within 2-week window after the abnormal TSH test
Time Frame: From first dose to 30 days post last dose (Up to 66 months)
Population: All treated participants with at least one on-treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 101 | 18
Participants
  TSH > ULN | 33 | 2
  TSH > ULN WITH TSH <= ULN AT BASELINE | 26 | 2
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN | 10 | 0
  TSH > ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 4 | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 23 | 0
  TSH < LLN | 38 | 5
  TSH < LLN WITH TSH >= LLN AT BASELINE | 37 | 4
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 7 | 0
  TSH < LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 2 | 1
  TSH < LLN WITH FT3/FT4 TEST MISSING | 15 | 2

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose (Up to 68 months)
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 29/101 | 10/18
Serious Adverse Events (participants affected / at risk) | 50/101 | 14/18
Other Adverse Events (participants affected / at risk) | 97/101 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=101) | Cohort B (N=18)
WARM TYPE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 0
MYOCARDITIS (Cardiac disorders) | 1 | 0
ADRENAL INSUFFICIENCY (Endocrine disorders) | 4 | 0
HYPERTHYROIDISM (Endocrine disorders) | 3 | 0
HYPOPHYSITIS (Endocrine disorders) | 6 | 0
VISION BLURRED (Eye disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 5 | 1
DIARRHOEA (Gastrointestinal disorders) | 6 | 1
DUODENITIS (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
IMMUNE-MEDIATED PANCREATITIS (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 4 | 1
DEATH (General disorders) | 1 | 0
FATIGUE (General disorders) | 2 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PYREXIA (General disorders) | 4 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 1 | 0
BACILLUS INFECTION (Infections and infestations) | 0 | 1
CELLULITIS ORBITAL (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1
MENINGITIS BACTERIAL (Infections and infestations) | 0 | 1
ORBITAL INFECTION (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 1
RASH PUSTULAR (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SYNOVIAL RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7 | 0
AMYLASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 | 0
LIPASE INCREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
INTRACRANIAL TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 9
TUMOUR PSEUDOPROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRAIN OEDEMA (Nervous system disorders) | 3 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
DYSAESTHESIA (Nervous system disorders) | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 3 | 0
HEADACHE (Nervous system disorders) | 1 | 0
HEMIPARESIS (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0
LACUNAR INFARCTION (Nervous system disorders) | 1 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0
PARTIAL SEIZURES (Nervous system disorders) | 0 | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 | 0
PRESYNCOPE (Nervous system disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 3 | 1
SYNCOPE (Nervous system disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 | 0
IMMUNE-MEDIATED NEPHRITIS (Renal and urinary disorders) | 1 | 0
NEPHRITIS (Renal and urinary disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
GRANULOMATOUS PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 4 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0
EMBOLISM (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=101) | Cohort B (N=18)
ANAEMIA (Blood and lymphatic system disorders) | 16 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 6 | 1
TACHYCARDIA (Cardiac disorders) | 4 | 1
EAR PAIN (Ear and labyrinth disorders) | 1 | 2
TINNITUS (Ear and labyrinth disorders) | 3 | 1
ADRENAL INSUFFICIENCY (Endocrine disorders) | 10 | 0
HYPERTHYROIDISM (Endocrine disorders) | 14 | 0
HYPOGONADISM (Endocrine disorders) | 0 | 1
HYPOPHYSITIS (Endocrine disorders) | 11 | 2
HYPOTHYROIDISM (Endocrine disorders) | 26 | 1
THYROIDITIS (Endocrine disorders) | 4 | 1
IRITIS (Eye disorders) | 0 | 2
OCULAR HYPERAEMIA (Eye disorders) | 2 | 1
PHOTOPHOBIA (Eye disorders) | 2 | 1
PHOTOPSIA (Eye disorders) | 2 | 2
VISION BLURRED (Eye disorders) | 14 | 5
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 1
VISUAL IMPAIRMENT (Eye disorders) | 4 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 5 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8 | 0
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 2 | 1
APHTHOUS ULCER (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 14 | 3
DIARRHOEA (Gastrointestinal disorders) | 51 | 8
DRY MOUTH (Gastrointestinal disorders) | 9 | 1
DYSPEPSIA (Gastrointestinal disorders) | 8 | 0
FLATULENCE (Gastrointestinal disorders) | 4 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 1
NAUSEA (Gastrointestinal disorders) | 53 | 10
ORAL DISORDER (Gastrointestinal disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 5 | 2
VOMITING (Gastrointestinal disorders) | 28 | 6
ASTHENIA (General disorders) | 2 | 1
CHILLS (General disorders) | 15 | 3
DISEASE PROGRESSION (General disorders) | 0 | 1
FATIGUE (General disorders) | 69 | 8
GAIT DISTURBANCE (General disorders) | 2 | 2
INFLUENZA LIKE ILLNESS (General disorders) | 13 | 1
LOCALISED OEDEMA (General disorders) | 1 | 1
MALAISE (General disorders) | 4 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 3 | 1
OEDEMA (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 18 | 3
PAIN (General disorders) | 5 | 1
PYREXIA (General disorders) | 28 | 4
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 2 | 1
CRYPTOCOCCAL FUNGAEMIA (Infections and infestations) | 0 | 1
IMPETIGO (Infections and infestations) | 0 | 1
ORAL CANDIDIASIS (Infections and infestations) | 6 | 1
SINUSITIS (Infections and infestations) | 8 | 1
TINEA CRURIS (Infections and infestations) | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 1
URINARY TRACT INFECTION (Infections and infestations) | 8 | 1
ESCHAR (Injury, poisoning and procedural complications) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 3 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 41 | 6
AMYLASE INCREASED (Investigations) | 17 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 39 | 3
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 12 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 7 | 1
BLOOD CREATININE INCREASED (Investigations) | 7 | 2
LIPASE INCREASED (Investigations) | 25 | 1
LIVER FUNCTION TEST INCREASED (Investigations) | 2 | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 8 | 1
PLATELET COUNT DECREASED (Investigations) | 9 | 0
WEIGHT DECREASED (Investigations) | 15 | 2
WEIGHT INCREASED (Investigations) | 7 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 6 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 30 | 4
DEHYDRATION (Metabolism and nutrition disorders) | 11 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 11 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 9 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 7 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 15 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 9 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 14 | 4
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 5 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 36 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 19 | 4
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 11 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 17 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 1
TUMOUR PSEUDOPROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
AMNESIA (Nervous system disorders) | 1 | 1
APHASIA (Nervous system disorders) | 6 | 3
ATAXIA (Nervous system disorders) | 2 | 1
BALANCE DISORDER (Nervous system disorders) | 0 | 1
COORDINATION ABNORMAL (Nervous system disorders) | 1 | 1
DIZZINESS (Nervous system disorders) | 18 | 4
DYSARTHRIA (Nervous system disorders) | 0 | 1
DYSGEUSIA (Nervous system disorders) | 7 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 4 | 1
HEADACHE (Nervous system disorders) | 52 | 8
HYPOAESTHESIA (Nervous system disorders) | 4 | 1
LETHARGY (Nervous system disorders) | 1 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 2 | 1
PARAESTHESIA (Nervous system disorders) | 11 | 1
PAROSMIA (Nervous system disorders) | 0 | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 7 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 1
SEIZURE (Nervous system disorders) | 3 | 2
SYNCOPE (Nervous system disorders) | 4 | 2
ANXIETY (Psychiatric disorders) | 5 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 7 | 3
DEPRESSION (Psychiatric disorders) | 6 | 1
INSOMNIA (Psychiatric disorders) | 23 | 5
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | 1
NEPHRITIS (Renal and urinary disorders) | 0 | 1
NOCTURIA (Renal and urinary disorders) | 2 | 1
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 33 | 6
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
INCREASED BRONCHIAL SECRETION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 15 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 9 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 5 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 10 | 3
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 6 | 1
MACULE (Skin and subcutaneous tissue disorders) | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 6 | 0
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 0 | 1
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 42 | 4
RASH (Skin and subcutaneous tissue disorders) | 14 | 3
RASH MACULAR (Skin and subcutaneous tissue disorders) | 3 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 42 | 5
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 5 | 2
SKIN HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 10 | 1
VITILIGO (Skin and subcutaneous tissue disorders) | 7 | 0
HOT FLUSH (Vascular disorders) | 5 | 1
HYPERTENSION (Vascular disorders) | 13 | 0
HYPOTENSION (Vascular disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT02320058/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT02320058/SAP_001.pdf